CLINICAL TRIAL: NCT01124318
Title: Phase II Double Blind Placebo-controled Randomized Comparative Multicentered Study of Efficacy and Safety of Lactofiltrum, Orally Administered Tablets (Produced by AVVA RUS, JSC) to Treat Atopic Dermatitis in Adults
Brief Title: A Pilot Study of Lactofiltrum to Treat Atopic Dermatitis in Adults
Acronym: LF-AD-09
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Avva Rus, JSC (Industry)
Collaborators: Moscow State University of Medicine and Dentistry (Other); Moscow Dermatovenerologic Clinical Dispensary № 1 (Unknown)
Responsible Party: Prof. Yuriy Perlamutrov, Head of dermatovenerologic diseases department, Moscow State University of Medicine and Dentistry
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04/09-AVVA RUS
Record Dates: First submitted 2010-04-28; First posted 2010-05-17 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Atopic Dermatitis
Keywords: Lactofiltrum; atopic dermatitis; itching; Dermatological Index of Life Quality; SCORAD; Behavioral Rating Scores
MeSH Terms: conditions — Dermatitis, Atopic; Pruritus | interventions — Lactulose; Lignin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactofiltrum (Active Comparator)
  Interventions: Drug: Lactofiltrum
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lactofiltrum — Lactofiltrum (hydrolytic lignin 0.355, lactulose 0.12) 2 tablets three times a day before meals during 21 days
  Other Names: Lactulose; Lignin
  Arms: Lactofiltrum
Drug: Placebo — Placebo 2 tablets 3 times a day before meals during 21 days
  Arms: Placebo

SUMMARY:
The purpose is to study efficacy of Lactofiltrum in adult patients with atopic dermatitis. Lactofiltrum consists of 85% of hidrolytic lignin and 15% of lactulose and acts as an enterosorbent, which enables to enhance metabolism and elimination of endotoxins and to normalize metabolic and immune processes. Additionally, lactulose stimulates Bifidobacterium flora and in aggregate it could improve skin condition afflicted by atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-60 y.o. diagnosed with atopic dermatitis according to the UK refinement of the Hanifin-Rajka diagnostic criteria;
* SCORAD Index more than 25.

Exclusion Criteria:

* pregnancy and breast-feeding;
* severe diseases;
* concomitant infection diseases (including parasitic ones);
* diffusive connective-tissue (autoimmune) diseases;
* renal and hepatic failure;
* systemic or topical treatment with antibiotics, steroids, immunosuppressive, cytostatic or antimetabolite agents by the time of inclusion into the study;
* concomitant skin diseases: skin lymphoma, scab, lichen ruber planus, psoriasis;
* professional activity involving skin injury, exposure to cold, insolation, ultraviolet radiation;
* psychoses;
* application of pre-, probiotics, antibiotics, neuroleptics or tranquilizers 2 weeks before inclusion or during participation in the study;
* participation in other clinical study 1 month before inclusion or during participation in the proposed study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
SCORAD Index | Day 21 after start of the intervention
  The Scoring of Atopic Dermatitis (SCORAD) index is a composite index (0-100 scores) measured by blinded physician assessing three main clinical features of the disease (separate scales), namely area of lesion, clinical severity, subjective symptoms.

SECONDARY OUTCOMES:
SCORAD Index | Day 30 after end of the intervention
  The Scoring of Atopic Dermatitis (SCORAD) index is a composite index (0-100 scores) measured by blinded physician assessing three main clinical features of the disease (separate scales), namely area of lesion, clinical severity, subjective symptoms.
SCORAD Index | Day 10 after start of the intervention
  The Scoring of Atopic Dermatitis (SCORAD) index is a composite index (0-100 scores) measured by blinded physician assessing three main clinical features of the disease (separate scales), namely area of lesion, clinical severity, subjective symptoms.
Dermatological Index of Life Quality | Day 10 after start of the intervention
  The Dermatological Index of Life Quality is a index (0-30 scores) representing patient's life quality deteriorations related to a skin disease (self-reported questionnaire).
Dermatological Index of Life Quality | Day 21 after start of the intervention
  The Dermatological Index of Life Quality is a index (0-30 scores) representing patient's life quality deteriorations related to a skin disease (self-reported questionnaire).
Dermatological Index of Life Quality | Day 30 after end of the intervention
  The Dermatological Index of Life Quality is a index (0-30 scores) representing patient's life quality deteriorations related to a skin disease (self-reported questionnaire).
BRS Index | Day 10 after start of the intervention
  Behavioral rating scores (BRS) measures severity of itching.
BRS Index | Day 21 after start of the intervention
  Behavioral rating scores (BRS) measures severity of itching.
BRS Index | Day 30 after end of the intervention
  Behavioral rating scores (BRS) measures severity of itching.
Blood test | Day 21 after start of the intervention
  It includes routine blood cells' counting and measurement of erythrocyte sedimentation rate and serum concentration of hemoglobin.
Biochemical blood analysis | Day 21 after start of the intervention
  It includes routine measurements of serum concentrations of biochemical compounds including proteins, glucose, enzymes, creatinine, urea, potassium, sodium, bilirubin.
Urine analysis | Day 21 after start of the intervention
  It includes routine measurements of urine concentrations of biochemical compounds including proteins and glucose, counting of cells, detection of bacteria and urinometry.

CONTACTS AND LOCATIONS:
Overall Officials: Yuriy Perlamutrov, MD, DrSc, Principal Investigator — Moscow State University of Medicine and Dentistry; Nickolay A. Kryuchkov, MD, PhD, MPH, Study Director — Avva Rus, JSC; Lyudmila Kobeleva, MD, PhD, Study Director — Avva Rus, JSC
Locations (2):
- Russia (2):
  - Moscow Dermatovenerologic Clinical Dispensary № 1, Moscow, Moscow
  - Moscow State University of Medicine and Dentistry, Moscow, Moscow